CLINICAL TRIAL: NCT04737564
Title: Attachment and Biobehavioral Catch-up With Child Protective Services-Involved Parents: Testing Effectiveness in the Community
Brief Title: Boosting Infant Resilience and Development
Acronym: earlyBIRD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Stony Brook University (Other)
Collaborators: University of Delaware (Other)
Responsible Party: Principal Investigator, Kristin Bernard, Associate Professor, Stony Brook University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R01MH119310 (NIH)
Record Dates: First submitted 2021-01-15; First posted 2021-02-04 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-05

CONDITIONS: Child Maltreatment

STUDY DESIGN:
Intervention Model Description: The standard Attachment and Biobehavioral Catch-up intervention (ABC10) is a 10-session home-visiting intervention. The ABC parenting targets include: nurturing children when they are distressed (Sessions 1 and 2), following the child's lead in play (Sessions 3 and 4), and avoiding harsh or frightening behavior (Sessions 5 and 6). Sessions 7 and 8 help parents consider how their own experiences of being parented affect their sensitivity, and Sessions 9 and 10 consolidate gains with additional practice. Session content focusing on parenting targets is guided by a manual. Additionally, parent coaches make frequent "in-the-moment" comments (at least once per minute) about parent-child interactions as they occur in session, and use video feedback.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ABC10 + SEEK (Experimental): Participants assigned to this arm will receive the standard Attachment and Biobehavioral Catch-up intervention (ABC 10) as well as SEEK (Safe Environment for Every Kid).
  Interventions: Behavioral: Attachment and Biobehavioral Catch-up (ABC10); Behavioral: Safe Environment for Every Kid (SEEK)
- ABC3 + SEEK (Experimental): Participants assigned to this arm will receive an abbreviated version of the Attachment and Biobehavioral Catch-up intervention (ABC 3) as well as SEEK (Safe Environment for Every Kid).
  Interventions: Behavioral: Attachment and Biobehavioral Catch-up, Brief (ABC3); Behavioral: Safe Environment for Every Kid (SEEK)
- SEEK Only (Active Comparator): Participants assigned to this arm will receive SEEK (Safe Environment for Every Kid) only.
  Interventions: Behavioral: Safe Environment for Every Kid (SEEK)

INTERVENTIONS:
Behavioral: Attachment and Biobehavioral Catch-up (ABC10) — The ABC parenting targets include: nurturing children when they are distressed (Sessions 1 and 2), following the child's lead in play (Sessions 3 and 4), and avoiding harsh or frightening behavior (Sessions 5 and 6). Sessions 7 and 8 help parents consider how their own experiences of being parented affect their sensitivity, and Sessions 9 and 10 consolidate gains with additional practice. Session content focusing on parenting targets is guided by a manual. Additionally, parent coaches make frequent "in-the-moment" comments (at least once per minute) about parent-child interactions as they occur in session, and use video feedback.
  Arms: ABC10 + SEEK
Behavioral: Attachment and Biobehavioral Catch-up, Brief (ABC3) — The 3-session Attachment and Biobehavioral Catch-up intervention (ABC 3) is a brief version of the standard protocol. Parents who receive ABC 3 will receive the first 3 sessions of the ABC intervention, which focus on enhancing parental sensitivity (i.e., nurturance to distress, following the child's lead) by providing in-the-moment feedback on parent-child interactions, video feedback, and discussion of manualized content. ABC 3 was adapted from the standard protocol based on modeling of session-by-session data that demonstrated that, on average, most of the change in parental sensitivity happens in the first several sessions of the intervention.
  Arms: ABC3 + SEEK
Behavioral: Safe Environment for Every Kid (SEEK) — Safe Environment for Every Kid (SEEK) is an evidence-based screening and referral system to facilitate parents' access to services for risk factors for maltreatment, including: mental health, substance abuse, intimate partner violence, harsh parenting, major parental stress, and food insecurity. Parents first complete the SEEK Parent Questionnaire with the help of an outreach worker. Following the SEEK protocol, handouts will be provided that address the identified problems and parents will be referred to partnering organizations in the community. Any additional work is completed by phone. The developer of the intervention, Howard Dubowitz, is a consultant on this application and will provide support around effective implementation.

SUMMARY:
Childhood maltreatment represents an urgent public health problem, as it is highly prevalent, significantly increases risk for chronically impairing mental health problems, tends to persist across generations, and is very costly to society at large. Leveraging an existing partnership between a community-based organization and child welfare system, this project will examine the effectiveness of the Attachment and Biobehavioral Catch-up (ABC) intervention, which targets sensitivity among parents who have maltreated their children. Findings will have substantial public health impact by assessing the effectiveness of the ABC intervention in a community context, identifying modifiable mechanistic pathways by which the ABC intervention may prevent later mental health problems, and identifying treatment moderators that may promote more targeted, cost-effective approaches to prevention.

DETAILED DESCRIPTION:
This effectiveness trial leverages an existing partnership between Power of Two, a non-profit organization in New York City (NYC) that delivers the ABC intervention to infants with child welfare involvement; NYC's Administration for Children Services (ACS) that oversees the child welfare system; and ACS-contracted preventive agencies that refer families to Power of Two. We will assess the effectiveness of the ABC intervention in engaging parental sensitivity, the intervention mechanism, using a multi-method approach (behavioral observation, neural activity via event-related potentials [ERP]), and in enhancing child outcomes; we will assess whether the purported intervention mechanism mediates the association between the intervention and child outcomes; and we will examine moderators of treatment effectiveness that could allow personalizing the intervention to individual needs. Participants will include 360 parents and their 6- to 24-month-old infants with indicated reports of maltreatment. Parents will be randomized to one of three conditions: an evidence-based screen-and-refer intervention (Safe Environment for Every Child [SEEK]16), SEEK plus the first three sessions of ABC (ABC 3), or SEEK plus the standard ABC protocol (ABC 10). Parents and their young children will be assessed at intake, after ABC session 3 (or equivalent for SEEK only condition), and at 6 and 12 months post-intake. Parental sensitivity and child functioning will be assessed at each time-point, and parental neural activity will be assessed at intake and 6 months post-intake.

The proposed research will address the following aims:

Aim 1: Examine effectiveness of the ABC intervention in a community context.

1a. Examine whether the ABC intervention engages the treatment mechanism. Parents randomized to ABC 10 are expected to show greater gains in observed sensitivity than parents randomized to SEEK.

1b. Examine whether ABC enhances parental neural activity. Parents randomized to ABC 10 are expected to show greater gains in neural activity associated with sensitivity than parents randomized to SEEK.

1. c. Examine whether the ABC intervention affects child outcomes. Children of parents randomized to ABC 10 are expected to show lower rates of disorganized attachment, more normative cortisol production, and less behavioral dysregulation than children of parents randomized to SEEK.

   Aim 2: Examine mediation effects.
2. a. Examine the extent to which target engagement leads to changes in child outcomes. Changes in parental sensitivity are expected to mediate the association between intervention participation and child outcomes.

2b. Examine whether changes in parental neural activity are key for sustained change in parental sensitivity. Changes in parental neural activity are expected to mediate the association between intervention participation and parental sensitivity.

Aim 3 (Exploratory): Examine moderation effects. Examine whether cumulative risk moderates intervention effects. More specifically, we will explore whether parents with lower cumulative risk indices respond more favorably to ABC 3 than parents with higher cumulative risk indices, whereas those with higher cumulative risk indices require the full ABC 10 protocol. We will also examine other variables, such as child sex, as possible moderators.

ELIGIBILITY:
Inclusion Criteria:

* Have an open preventive case following an indicated report of maltreatment (to be confirmed by referring agency)
* Reside in Brooklyn or the Bronx
* Be the biological parent and primary caregiver of a child between 6 and 24 months old, and - Identify English or Spanish as their preferred language.

Exclusion Criteria:

- None

Ages: 6 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 360 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Parental sensitivity | Approximately 4 weeks post-intake (After ABC Session 3 or the equivalent for SEEK only dyads)
  After ABC Session 3 (or the equivalent for SEEK only dyads), parental sensitivity will be coded on the basis of a 30-minute semi-structured interaction, including a play task and challenge/ distress tasks. The parent will be given 3 bags of toys and asked to play with the toys in each of the three bags in order and complete a series of challenge/distress-eliciting tasks that vary based on child age, such as changing the child's clothes, withholding an attractive toy, and completing research measures while the child is present. We will use the NICHD SECCYD methods for coding parental sensitivity, including scales for sensitivity to distress (consistent with the ABC target of nurturance), sensitivity to non-distress (consistent with the ABC target of following the child's lead), and positive regard (consistent with the ABC target of delight). Raters will be trained to better than 85% inter-rater reliability and reliability will be carefully monitored, with all assessments double-coded.
Parental sensitivity | At 6-months post-intake
  At 6 months post-intake (or the equivalent for SEEK only dyads), parental sensitivity will be coded on the basis of a 30-minute semi-structured interaction, including a play task and challenge/ distress tasks. The parent will be given 3 bags of toys and asked to play with the toys in each of the three bags in order and complete a series of challenge/distress-eliciting tasks that vary based on child age, such as changing the child's clothes, withholding an attractive toy, and completing research measures while the child is present. We will use the NICHD SECCYD methods for coding parental sensitivity, including scales for sensitivity to distress, sensitivity to non-distress, and positive regard. Raters will be trained to better than 85% inter-rater reliability and reliability will be carefully monitored, with all assessments double-coded.
Parental sensitivity | At 12-months post-intake
  At 12 months post-intake (or the equivalent for SEEK only dyads), parental sensitivity will be coded on the basis of a 30-minute semi-structured interaction, including a play task and challenge/ distress tasks. The parent will be given 3 bags of toys and asked to play with the toys in each of the three bags in order and complete a series of challenge/distress-eliciting tasks that vary based on child age, such as changing the child's clothes, withholding an attractive toy, and completing research measures while the child is present. We will use the NICHD SECCYD methods for coding parental sensitivity, including scales for sensitivity to distress, sensitivity to non-distress, and positive regard. Raters will be trained to better than 85% inter-rater reliability and reliability will be carefully monitored, with all assessments double-coded.
Parental neural activity: N170 to emotional faces | 6 months post-intake
  At 6 months post-intake, parental neural activity will be assessed using an event-related potential (ERP) task. Parents will categorize photographs of infants with different emotional expressions (crying, laughing, neutral), while continuous EEG is recorded (Bernard et al., 2015). The N170 (an early perceptual ERP component that indexes processing of faces) will be measured as the average amplitude within a time window of 140 to 180 ms at electrodes P7 and P8. After data processing (re-referencing, artifact rejection), residualized difference scores will be computed that reflect the magnitude of the difference in N170 responses to emotional faces versus neutral faces.
Parental neural activity: Late positive potential (LPP) to emotional faces | 6 months post-intake
  At 6 months post-intake, parental neural activity will be assessed using an event-related potential (ERP) task. Parents will categorize photographs of infants with different emotional expressions (crying, laughing, neutral), while continuous EEG is recorded (Bernard et al., 2015). The late positive potential (LPP; a late ERP component that indexes sustained attention and evaluation of emotionally-salient stimuli) will be measured as the average amplitude at the Pz electrode from 300 to 650 ms post-stimulus. After data processing (re-referencing, artifact rejection), residualized difference scores will be computed that reflect the magnitude of the difference in LPP responses to emotional faces versus neutral faces.
Child attachment | 6 months post-intake
  At 6 months post-intake, the Strange Situation procedure (Ainsworth et al., 1978) will be conducted. The Strange Situation consists of a series of episodes including two 3-minute separations, each followed by 3-minute reunions. The child's behavior upon reunion with the parent is coded for continuous scales (i.e., proximity seeking, contact maintenance, avoidance, resistance) and children are classified as secure, insecure-avoidant, or insecure-resistant. Following the Main & Solomon (1990) system, disorganized attachment behavior is also coded on a continuous scale, and children may receive a primary classification of disorganized attachment. Elizabeth Carlson, an expert coder, will serve as a consultant on this project and complete reliability coding for 25% of videos.
Child diurnal cortisol rhythm at 6 months post-intake | 6 months post-intake
  At 6 months post-intake, children's diurnal cortisol rhythms will be assessed. Cortisol is an end product of the hypothalamic-pituitary-adrenal (HPA) axis. The normative pattern is a high wake-up level, decreasing throughout the day, with the nadir in the evening. Parents will collect child saliva samples by rubbing an oral swab in the child's mouth at wake-up (morning) and bedtime (evening) for 3 consecutive days. Saliva samples will be assayed using the Salimetrics, Inc. High Sensitivity Salivary Cortisol Enzyme Immunoassay Kit. All samples from a child at a single time-point will be run in duplicate on the same assay plate, along with a control. Cortisol values, measured in ?g/dl, will be log-transformed. We will examine changes in the diurnal rhythm (i.e., slope) from wake-up to bedtime.
Child diurnal cortisol rhythm at 12 months post-intake | 12 months post-intake
  At 12 months post-intake, children's diurnal cortisol rhythms will be assessed. Cortisol is an end product of the hypothalamic-pituitary-adrenal (HPA) axis. The normative pattern is a high wake-up level, decreasing throughout the day, with the nadir in the evening. Parents will collect child saliva samples by rubbing an oral swab in the child's mouth at wake-up (morning) and bedtime (evening) for 3 consecutive days. Saliva samples will be assayed using the Salimetrics, Inc. High Sensitivity Salivary Cortisol Enzyme Immunoassay Kit. All samples from a child at a single time-point will be run in duplicate on the same assay plate, along with a control. Cortisol values, measured in ?g/dl, will be log-transformed. We will examine changes in the diurnal rhythm (i.e., slope) from wake-up to bedtime.
Child behavior regulation (Infant Externalizing Questionnaire) after ABC session 3 (or equivalent) | Approximately 4 weeks post-intake (After ABC Session 3 or the equivalent for SEEK only dyads)
  After ABC Session 3 (or the equivalent for SEEK-only dyads), parents will complete the Infant Externalizing Questionnaire (IEQ; Lorber et al., 2017) when children are 24 months of age or younger. The IEQ is a measure of infant aggression (7 items) and defiance (4 items) and shows good internal consistency, longitudinal stability, interparental agreement, and concurrent and predictive validity.
Child behavior regulation (Infant Externalizing Questionnaire) at 6 months post-intake | 6 months post-intake
  At 6 months post-intake, parents will complete the Infant Externalizing Questionnaire (IEQ; Lorber et al., 2017) when children are 24 months of age or younger. The IEQ is a measure of infant aggression (7 items) and defiance (4 items) and shows good internal consistency, longitudinal stability, interparental agreement, and concurrent and predictive validity.
Child behavior regulation (Infant Externalizing Questionnaire) at 12 months post-intake | 12 months post-intake
  At 12 months post-intake, parents will complete the Infant Externalizing Questionnaire (IEQ; Lorber et al., 2017) when children are 24 months of age or younger. The IEQ is a measure of infant aggression (7 items) and defiance (4 items) and shows good internal consistency, longitudinal stability, interparental agreement, and concurrent and predictive validity.
Child behavior regulation (Child Behavior Checklist) at 6 months post-intake | 6 months post-intake
  At 6 months post-intake, parents will complete the Child Behavior Checklist 1? - 5 (CBCL; Achenbach & Rescorla, 2001) for children at least 18 months old, which will allow us to assess both internalizing and externalizing behaviors. The use of the IEQ and the CBCL at overlapping waves of data collection is intentional because it allows us to correct for switching indicators in statistical analyses.
Child behavior regulation (Child Behavior Checklist) at 12 months post-intake | 12 months post-intake
  At 12 months post-intake, parents will complete the Child Behavior Checklist 1? - 5 (CBCL; Achenbach & Rescorla, 2001), which will allow us to assess both internalizing and externalizing behaviors. The use of the IEQ and the CBCL at overlapping waves of data collection is intentional because it allows us to correct for switching indicators in statistical analyses.
Child behavior regulation (Disruptive Behavior Diagnostic Observation Schedule) at 6 months post-intake | 6 months post-intake
  At the 6 months post-intake assessment, the Disruptive Behavior Diagnostic Observation Schedule (DB-DOS; Wakschlag et al., 2008) will be administered. The DB-DOS is an observational assessment that involves a series of "presses" that challenge children's emotional and behavioral regulatory capacities; the DB-DOS demonstrates good reliability and validity. Given that children will be between 12 and 30 months at the 6 months post-intake time-point, we will administer the infant/toddler DB-DOS protocol, which allows for the assessment of child irritability and frustration, key behavioral regulation constructs that are predictive of later difficulties with disruptive behavior disorders.

SECONDARY OUTCOMES:
Client satisfaction with services after ABC Session 3 (or equivalent) | Approximately 4 weeks post-intake (After ABC Session 3 or the equivalent for SEEK only dyads)
  After ABC Session 3 (or the equivalent for SEEK-only dyads), client satisfaction with services will be assessed with the Client Satisfaction Questionnaire (CSQ-8; Larson et al., 1979). The CSQ-8 is an 8-item questionnaire that asks participants about their satisfaction with services received (e.g., to what extent services met needs, likelihood of recommending a friend). The CSQ-8 provides a good measure of participants' perception of services received.
Client satisfaction with services at 6 months post-intake | 6 months post-intake
  At 6 months post-intake, client satisfaction with services will be assessed with the Client Satisfaction Questionnaire (CSQ-8; Larson et al., 1979). The CSQ-8 is an 8-item questionnaire that asks participants about their satisfaction with services received (e.g., to what extent services met needs, likelihood of recommending a friend). The CSQ-8 provides a good measure of participants' perception of services received.
Child maltreatment after ABC Session 3 (or equivalent) | Approximately 4 weeks post-intake (After ABC Session 3 or the equivalent for SEEK only dyads)
  After ABC Session 3 (or the equivalent for SEEK-only dyads), we will assess subsequent reports of maltreatment to ACS, which will be coded as reported, investigated, and substantiated. In addition, we will code available records using the Modified Maltreatment Classification System (Barnett et al., 1993) for type and severity of maltreatment exposure.
Child maltreatment at 6 months post-intake | 6 months post-intake
  At 6 months post-intake, we will assess subsequent reports of maltreatment to ACS, which will be coded as reported, investigated, and substantiated. In addition, we will code available records using the Modified Maltreatment Classification System (Barnett et al., 1993) for type and severity of maltreatment exposure.
Child maltreatment at 12 months post-intake | 12 months post-intake
  At 12 months post-intake, we will assess subsequent reports of maltreatment to ACS, which will be coded as reported, investigated, and substantiated. In addition, we will code available records using the Modified Maltreatment Classification System (Barnett et al., 1993) for type and severity of maltreatment exposure.

IPD SHARING:
Plan to Share IPD: Undecided